CLINICAL TRIAL: NCT00294645
Title: Pacemaker Remote Follow-up Evaluation and Review
Brief Title: PREFER (Pacemaker Remote Follow-Up Evaluation and Review)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Medtronic, Cardiac Rhythm Disease Management Clinical Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 701
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Results first posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Bradycardia; Arrhythmia
Keywords: Remote Follow Up; Diagnostic; Bradycardia
MeSH Terms: conditions — Bradycardia; Arrhythmias, Cardiac; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Transtelephonic monitoring at 2 month intervals
  Interventions: Other: Transtelephonic monitoring (TTM)
- Remote (Active Comparator): Medtronic CareLink® Network remote pacemaker interrogation at 3 month intervals
  Interventions: Other: Medtronic CareLink® Network

INTERVENTIONS:
Other: Transtelephonic monitoring (TTM) — TTM conducted at 2 month intervals. For patients with dual-chamber pacemakers, an in-office visit was required at 6 months (rather than TTM transmission for patients with single-chamber pacemakers). Follow-up frequency established to mimic best case standard of care when utilizing TTM for follow-up. A 12-month in-office visit completed the follow-up period.
  Arms: Control
Other: Medtronic CareLink® Network — Remote pacemaker interrogation conducted at 3 month intervals. Follow-up frequency established to mimic best case standard of care when utilizing implantable cardioverter defibrillator (ICD) remote interrogation for follow-up. A 12-month in-office visit completed the follow-up period.
  Arms: Remote

SUMMARY:
The purpose of the study is to compare remote pacemaker follow-up to current standard of care follow-up. The study will compare the rate of first diagnosis of clinically actionable events between patients who utilize the Medtronic Carelink® Network (Remote arm) versus patients who are followed via routine office visits augmented by transtelephonic monitoring (TTM)(Control arm).

DETAILED DESCRIPTION:
The Clinically Actionable Events (CAE) were identified based on their relation to other comorbidities that may increase the risk of a serious cardiac event. The defined events are:

1. Atrial Tachycardia/Atrial Fibrillation (AT/AF) episodes of greater than 48 hours defined as two consecutive days in which the device records at least 18 hours of AT/AF per day
2. Ventricular pacing that has increased by 30 percent (relative) since the last device interrogation
3. A sensed ventricular response of greater than 100 beats per minute (BPM) during atrial tachyarrhythmia for at least 20 percent of the time since the previous device interrogation
4. Runs of non-sustained ventricular tachycardia (NSVT) greater than 5 beats
5. New onset of AT/AF among patients with no history of AT/AF
6. Loss of atrial capture
7. Loss of ventricular capture
8. Increase in atrial pacing voltage threshold greater than 1 volt (V)
9. Increase in ventricular pacing voltage threshold greater than 1 volt (V)
10. & 11. Significant change in atrial or ventricular lead impedance, defined as any of the following:

    1. Less than 200 or greater than 2000 ohms (Ω)
    2. Unstable lead impedance deemed to be clinically actionable
    3. Greater than 50 percent change in lead impedance since last interrogation

12. Elective Replacement Indicator (ERI)/Battery End of Life (EOL) indicators

ELIGIBILITY:
Inclusion Criteria:

* Patient has been previously implanted with a dual-chamber or single-chamber EnPulse®, Kappa 900®, or Adapta® device
* Patient agrees to complete all required follow-up transmissions and in-office visits
* Patient is capable of operating the TTM monitor and Medtronic CareLink monitor

Exclusion Criteria:

* Patient is an immediate candidate for an implantable cardioverter defibrillator (ICD)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 980 (Actual)
Dates: Start 2004-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PREFER Study Team, Study Chair — Medtronic
Locations (45):
- United States (45):
  - Scottsdale, Arizona
  - Little Rock, Arkansas
  - Washington D.C., District of Columbia
  - Ormond Beach, Florida
  - Safety Harbor, Florida
  - Springfield, Illinois
  - Des Moines, Iowa
  - Lafayette, Louisiana
  - Bangor, Maine
  - Glen Burnie, Maryland
  - Takoma Park, Maryland
  - Burlington, Massachusetts
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - Hattiesburg, Mississippi
  - Jackson, Mississippi
  - Kansas City, Missouri
  - St Louis, Missouri
  - Great Falls, Montana
  - Omaha, Nebraska
  - Reno, Nevada
  - Ocean City, New Jersey
  - Paterson, New Jersey
  - Towaco, New Jersey
  - Voorhees Township, New Jersey
  - Mineola, New York
  - Raleigh, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Marion, Ohio
  - Tulsa, Oklahoma
  - Bend, Oregon
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Wynnewood, Pennsylvania
  - Columbia, South Carolina
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Corpus Christi, Texas
  - Houston, Texas
  - Plano, Texas
  - Temple, Texas
  - Tacoma, Washington
  - Wauwatosa, Wisconsin

REFERENCES:
- [Background] Chen J, Wilkoff BL, Choucair W, Cohen TJ, Crossley GH, Johnson WB, Mongeon LR, Serwer GA, Sherfesee L. Design of the Pacemaker REmote Follow-up Evaluation and Review (PREFER) trial to assess the clinical value of the remote pacemaker interrogation in the management of pacemaker patients. Trials. 2008 Apr 3;9:18. doi: 10.1186/1745-6215-9-18. PMID 18387185
- [Derived] Crossley GH, Chen J, Choucair W, Cohen TJ, Gohn DC, Johnson WB, Kennedy EE, Mongeon LR, Serwer GA, Qiao H, Wilkoff BL; PREFER Study Investigators. Clinical benefits of remote versus transtelephonic monitoring of implanted pacemakers. J Am Coll Cardiol. 2009 Nov 24;54(22):2012-9. doi: 10.1016/j.jacc.2009.10.001. PMID 19926006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from May 24, 2004 through March 30, 2007 at cardiology and electrophysiology clinics in the United States.
Pre-assignment Details: Of the 980 patients enrolled, 83 were excluded from analysis: incomplete informed consent forms (n=8), devices incompatible with the Medtronic CareLink® Network (n=7), from research centers that closed prior to cleaning data to the extent necessary for inclusion in cohort (n=67), and exited prior to Baseline assessment (n=1).
Groups:
- Standard of Care With TTM: Pacemaker patients followed by transtelephonic monitoring at 2 month intervals
- Remote Pacemaker Interrogation: Pacemaker patients followed by remote pacemaker interrogation at 3 month intervals
Period: Overall Study
Arm/Group | Standard of Care With TTM | Remote Pacemaker Interrogation
Started | 295 | 602
Completed | 247 | 510
Not Completed | 48 | 92
Not completed — Death | 10 | 18
Not completed — Lost to Follow-up | 1 | 10
Not completed — Withdrawal by Subject | 18 | 34
Not completed — Physician Decision | 15 | 20
Not completed — Other | 4 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care With TTM | Remote Pacemaker Interrogation | Total
Number analyzed (Participants) | 295 | 602 | 897
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 16 | 25.0
  Between 18 and 65 years | 74 | 169 | 243.0
  >=65 years | 212 | 417 | 629.0
Age Continuous [Mean (Standard Deviation); unit: years] | 69 (16.9) | 68 (16.7) | 68 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 290 | 443.0
  Male | 142 | 312 | 454.0
Region of Enrollment [Number; unit: participants]
  United States | 295 | 602 | 897.0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With First Diagnosis of Clinically Actionable Events (CAE) at 12 Months
Description: Clinically Actionable Events (CAE) are 12 events that were identified based on their relation to other comorbidities that may increase the risk of a serious cardiac event. The CAEs consist of several arrhythmias and device performance parameters such as: Atrial Tachycardia/Atrial Fibrillation (AT/AF) and loss of capture.
Time Frame: One year post-enrollment
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care With TTM | Remote Pacemaker Interrogation
Number analyzed (Participants) | 295 | 602
Percentage of participants | 35 | 47
Statistical Analysis 1: Comparison: Standard of Care With TTM vs Remote Pacemaker Interrogation; Null hypothesis: control rate = remote rate; Test type: Superiority or Other; p < 0.0001, Modified Peto-Peto; A one-sided test was used

2. Secondary Outcome: Proportion of Actions Taken in Response to the Diagnosis of Clinically Actionable Events
Description: Actions categories include: Referral, Office Visit, Medication (Med) Change, Hospitalization, Emergency Room (ER) Visit, Device Reprogrammed, System Modification, Increase Monitoring, Other
Time Frame: One year post-enrollment
Measure: Number; unit: Total number actions/total number CAEs
Arm/Group | Standard of Care With TTM | Remote Pacemaker Interrogation
Number analyzed (Participants) | 295 | 602
Total number actions/total number CAEs
  Referral | 0.005 | 0.006
  Office Visit | 0.016 | 0.043
  Med Change | 0.053 | 0.05
  Hospitalization | 0 | 0.012
  ER Visit | 0 | 0.001
  Device Reprogrammed | 0.016 | 0.028
  System Modification | 0 | 0.009
  Increase Monitoring | 0.011 | 0.009
  Other | 0.047 | 0.031

3. Secondary Outcome: Percentage of Participants With First Diagnosis of New Onset Atrial Tachycardia/Atrial Fibrillation (AT/AF) at 12 Months
Description: Compare time to first diagnosis in Remote and Control arms
Time Frame: One year post-enrollment
Population: Only participants without a history of Atrial Tachycardia/Atrial Fibrillation were included in analysis of this objective.
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care With TTM | Remote Pacemaker Interrogation
Number analyzed (Participants) | 139 | 282
Percentage of participants | 8 | 15

4. Secondary Outcome: Percentage of Participants With First Diagnosis of Sensed Ventricular Rate Greater Than 100 Beats Per Minute (BPM) During Atrial Tachycardia/Atrial Fibrillation at 12 Months
Description: Compare time to diagnosis in Control and Remote arms
Time Frame: One year post-enrollment
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care With TTM | Remote Pacemaker Interrogation
Number analyzed (Participants) | 295 | 602
Percentage of participants | 9 | 12

5. Secondary Outcome: Percentage of Participants With First Diagnosis of Atrial Tachycardia/Atrial Fibrillation Greater Than 48 Hours at 12 Months
Description: Compare time to diagnosis in Control and Remote arms
Time Frame: One year post-enrollment
Population: Cohort was subset of full cohort excluding participants with single chamber devices, thus the variance in number analyzed vs other endpoint analyses.
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care With TTM | Remote Pacemaker Interrogation
Number analyzed (Participants) | 266 | 557
Percentage of participants | 9 | 10

6. Secondary Outcome: Percentage of Participants With First Diagnosis of Ventricular Pacing Increase Greater Than 30 Percent at 12 Months
Description: Compare time to first diagnosis in Control and Remote arms
Time Frame: One year post-enrollment
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care With TTM | Remote Pacemaker Interrogation
Number analyzed (Participants) | 295 | 602
Percentage of participants | 4 | 8

7. Secondary Outcome: Percentage of Participants With First Diagnosis of Non-sustained Ventricular Tachycardia at 12 Months
Description: Compare time to first diagnosis in Control and Remote arms
Time Frame: One year post-enrollment
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care With TTM | Remote Pacemaker Interrogation
Number analyzed (Participants) | 295 | 602
Percentage of participants | 21 | 26

8. Secondary Outcome: Percentage of Participants With First Diagnosis of Loss of Atrial Capture at 12 Months
Description: Compare time to first diagnosis in Control and Remote arms
Time Frame: One year post-enrollment
Population: Analysis used subset of full cohort excluding participants with single chamber devices, thus the variance in number analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care With TTM | Remote Pacemaker Interrogation
Number analyzed (Participants) | 266 | 557
Percentage of participants | 0 | 0

9. Secondary Outcome: Percentage of Participants With First Diagnosis of Loss of Ventricular Capture at 12 Months
Description: Compare time to first diagnosis in Remote and Control arms
Time Frame: One year post-enrollment
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care With TTM | Remote Pacemaker Interrogation
Number analyzed (Participants) | 295 | 602
Percentage of participants | 0 | 1

10. Secondary Outcome: Percentage of Participants With an Increase in Atrial Pacing Voltage Threshold Greater Than 1 Volt (V) at 12 Months
Description: Compare time to first diagnosis in Remote and Control arms
Time Frame: One year post-enrollment
Population: Cohort was subset of full cohort excluding participants with single chamber devices, thus the variance in number analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care With TTM | Remote Pacemaker Interrogation
Number analyzed (Participants) | 266 | 557
Percentage of participants | 0 | 1

11. Secondary Outcome: Percentage of Participants With an Increase in Ventricular Pacing Voltage Threshold Greater Than 1 Volt (V) at 12 Months
Description: Compare time to first diagnosis in Control and Remote arms
Time Frame: One year post-enrollment
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care With TTM | Remote Pacemaker Interrogation
Number analyzed (Participants) | 295 | 602
Percentage of participants | 1 | 1

12. Secondary Outcome: Percentage of Participants With First Diagnosis of Change in Atrial Lead Impedance at 12 Months
Description: Compare time to first diagnosis in Control and Remote arms
Time Frame: One year post-enrollment
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care With TTM | Remote Pacemaker Interrogation
Number analyzed (Participants) | 266 | 557
Percentage of participants | 0 | 0

13. Secondary Outcome: Percentage of Participants With First Diagnosis of Change in Ventricular Lead Impedance at 12 Months
Description: Compare time to first diagnosis in Control and Remote arms
Time Frame: One year post-enrollment
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care With TTM | Remote Pacemaker Interrogation
Number analyzed (Participants) | 295 | 602
Percentage of participants | 1 | 1

14. Secondary Outcome: Percentage of Participants With First Diagnosis of Elective Replacement Indicator/Battery End of Life (ERI/EOL) at 12 Months
Description: Compare time to first diagnosis in Control and Remote arms
Time Frame: One year post-enrollment
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care With TTM | Remote Pacemaker Interrogation
Number analyzed (Participants) | 295 | 602
Percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected for this protocol.
Arm/Group | Standard of Care With TTM | Remote Pacemaker Interrogation
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, contracts allow investigators ("PI") to publish per the publication strategy/Clinical Investigation Plan following Medtronic's review for (a) disclosure of confidential information ("CI"), and (b) selection and order of publications by the publications committee. Any such CI is deleted prior to publication/presentation. Medtronic may not otherwise censor/interfere with the publication. PIs may not publish single-site data until the main multi-site publication has occurred.